CLINICAL TRIAL: NCT02028533
Title: Chronic Intranasal Oxytocin as an Adjunct to Methadone Maintenance Treatment in Patients With Co-occuring Opioid Use Disorder and Cocaine Use: A 2-week Pilot Study
Brief Title: Cocaine Opioid Oxytocin Option - Limited
Acronym: COOOL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 13-12534
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Opioid Use Disorder; Cocaine Use Disorder
Keywords: addiction; oxytocin; tolerability
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients 1 (Active Comparator): Participants will receive intranasal oxytocin 40 International Units (IU).
  Interventions: Drug: Oxytocin
- Patients 2 (Placebo Comparator): Participants will receive 40 International Units of intranasal placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: oxytocin nasal spray, Syntocinon
  Arms: Patients 1
Drug: Placebo
  Other Names: placebo nasal spray
  Arms: Patients 2

SUMMARY:
This is a pilot feasibility study assessing the tolerability of chronic administration of intranasal oxytocin to patients receiving methadone at an opioid replacement clinic who are actively using cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a patient in the San Francisco General Hospital Opioid Treatment Outpatient Program
* Stable dose of methadone for at least the past two weeks
* At least one routine urine toxicology screen positive for cocaine in the past month

Exclusion Criteria:

* Positive urine pregnancy test
* Use of illicit drugs in the past month (with the exception of cocaine or cannabis)
* Currently meets Diagnostic and Statistical Manual-5 (DSM-V) criteria for severe major depressive disorder with suicidal thoughts or actions
* History of psychotic or moderate-severe alcohol use disorder as defined by DSM-V criteria
* Severe neuropsychological disorder, brain trauma, epilepsy
* Sensitivity to preservatives (in particular E 216, E 218 and chlorobutanol hemihydrate)
* Nasal obstruction, discharge, or bleeding
* Habitually drinks large volumes of water
* Taking testosterone, estrogen/progesterone supplement, or serotonin-1a receptor agonists/antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with non-serious and serious adverse events | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Stauffer, MD, Principal Investigator — University of California, San Francisco; Joshua Woolley, MD, PhD, Study Director — University of California, San Francisco
Locations (1):
- San Francisco General Hospital Opiate Treatment Outpatient Program, San Francisco, California, United States